CLINICAL TRIAL: NCT06138028
Title: The Prospective Study of Sintilimab Combination With Chemotherapy Sequential Radiotherapy for Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Sintilimab and Chemotherapy Sequential Radiotherapy in Advanced Esophageal Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY202306702
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — TP protocol; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined chemo-immuno-irradiation (Experimental): TP regimen plus PD-1 inhibitor for 4 cycles then irradiation and PD-1 inhibitor maintenance therapy for 13 cycles.
  Interventions: Drug: TP regimen (cis-platinum ; Tocetaxel ) combined with PD-1 inhibitors（Sintilimab）

INTERVENTIONS:
Drug: TP regimen (cis-platinum ; Tocetaxel ) combined with PD-1 inhibitors（Sintilimab） — TP regimen (cis-platinum ; Tocetaxel ) combined with PD-1 inhibitors（Sintilimab）for 4 cycles, then irradiation of the residual lesions for 50Gy/2Gy/25f. After complete irradiation, sintilimab is administered every 21 days a cycle for additional 13 cycles.

SUMMARY:
This is an investigator-initiated, single-arm, exploratory clinical study.The study population consisted of treatment naive advanced esophageal squamous cell carcinoma patients. The purpose of this study was to evaluate the efficacy and safety of immunotherapy combined with chemotherapy and residual lesions irradiation of esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Stage IV esophagus squamous cell carcinoma.
2. Expected survival time ≥3 months
3. Enrolled patients must have at least one measurable lesion conforming to the RECIST V1.1 definition.
4. Physical fitness ECOG score of 0 or 1
5. Organ function levels must meet the following requirements and meet the following standards:

A) Bone marrow function: absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet count ≥90×10^9/L, hemoglobin ≥90 g/L; B) Liver function: Total bilirubin TBIL≤1.5×ULN (total bilirubin ≤3×ULN in Subjects with Gilbert's syndrome, liver cancer or liver metastasis), AST and ALT ≤2.5×ULN in patients without liver metastasis, AST and ALT ≤5.0×ULN in patients with liver metastasis; C) Renal function: Creatinine (Cr) ≤1.5×ULN, or creatinine clearance (Ccr) ≥50 mL/min (according to Cockcroft and Gault formula); D) Urine routine / 24-hour protein quantification: qualitative urine protein ≤1+ (if qualitative urine protein ≥2+, 24 hours < 1g can be included); E) Cardiac function: left ventricular ejection fraction ≥50%; F) Coagulation function: International standardized ratio (INR) ≤1.5×ULN, and activated partial thrombin time (APTT) ≤1.5×ULN;

Exclusion Criteria:

1. Known or suspected history of active autoimmune diseases, autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitaritis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes)
2. Have a history of immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency disease, or history of organ transplantation and bone marrow transplantation；Interstitial lung disease, drug-induced pneumonia,requiring steroid therapy or active pneumonia with clinical symptoms or severe pulmonary dysfunction；
3. There are clinical symptoms or diseases of the heart that are not well controlled, such as: (1) heart failure of NYHA class 2 or higher (2) unstable angina (3) myocardial infarction within 24 weeks (4) clinical need for treatment or Interventional supraventricular or ventricular arrhythmia；
4. Have a tendency to hereditary bleeding or coagulopathy. Clinically significant bleeding symptoms or clear bleeding tendency within 3 months prior to enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood++ and above；
5. Allergic reactions to test drugs for this application；
6. Pregnant or lactating women； Those whom the investigator considered unsuitable for inclusion。

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 24 months
  time from enrollment to patients death
Progression-free survival (PFS) | up to 12 months
  time from disease progression or patient death

SECONDARY OUTCOMES:
overall response rate (ORR) | up to 12 weeks
  complete response plus partial response
toxicities | up to 12 weeks
  toxicities according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Qingdao Central Hospital, Qingdao Cancer Hospital, Qingdao, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong

IPD SHARING:
Plan to Share IPD: Undecided